CLINICAL TRIAL: NCT03714360
Title: The Effect of Tranexamic Acid on Duration of Surgery, Bleeding and Complications. A Double Blind, Placebo-controlled, Randomised Study of Patients Undergoing Elective Lumbar Spine Surgery.
Brief Title: The Effect of Tranexamic Acid. A Randomised Study of Patients Undergoing Elective Lumbar Spine Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mikkel Østerheden Andersen (Other)
Responsible Party: Sponsor-Investigator, Mikkel Østerheden Andersen, Professor, Spine Centre of Southern Denmark
Organization: Spine Centre of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-20150072
Record Dates: First submitted 2018-10-15; First posted 2018-10-22 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Pharmacological Action
Keywords: TXA;decompression; discectomy; operative time; blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXA tranexamic acid (Experimental): a single dose of 10 mg/kg of TXA, with a maximum dose of 1g. Administered as IV injection and marked as 'project-drug' and amount (mL) in the medical record.
  Interventions: Drug: Tranexamic Acid
- Sodium Chloride 0,9% (Placebo Comparator): an equivalent volume 0.9 % Sodium Chloride.
  Interventions: Drug: Sodium Chloride 0,9%

INTERVENTIONS:
Drug: Tranexamic Acid — patients with ASA(American Society of Anesthesiologists grades) 1 to 2, scheduled to undergo lumbar decompressive surgery at Middelfart Hospital. Patients were randomized, in blocks of 10, to two groups: TXA or placebo. Anticoagulation therapy was discontinued 2-7 days preoperatively. Prior to the incision, patients received either a bolus of TXA (10mg/kg), or an equivalent volume of saline solution (placebo).
  Other Names: TXA
  Arms: TXA tranexamic acid
Drug: Sodium Chloride 0,9% — Sodium Chloride 0,9%
  Arms: Sodium Chloride 0,9%

SUMMARY:
In this randomized double blind placebo controlled study of tranexamic acid during minor spinal surgery, mean postoperative blood loss in the patients who received TXA was statistically significantly lower compared to placebo.

DETAILED DESCRIPTION:
Study Design: Double-blind, randomized, placebo-controlled, parallel-group study.

Objective: To investigate the effect of tranexamic acid (TXA) compared to placebo in low-risk adult patients undergoing elective minor lumbar spine surgery on operative time, estimated blood loss and complications.

Summary of Background Data: Studies have shown that TXA reduces blood loss during major spine surgery. There are no studies on the effect of TXA in minor lumbar spine surgery on operative time, intraoperative and postoperative blood loss and complications.

Methods: We enrolled patients with ASA grades 1 to 2, scheduled to undergo lumbar decompressive surgery at Middelfart Hospital. Patients with thromboembolic disease, coagulopathy, hypersensitivity to TXA or history of convulsion were excluded. Patients were randomized, in blocks of 10, to two groups: TXA or placebo. Anticoagulation therapy was discontinued 2-7 days preoperatively. Prior to the incision, patients received either a bolus of TXA (10mg/kg), or an equivalent volume of saline solution (placebo).

ELIGIBILITY:
Inclusion Criteria:

* patients referred to the Centre for Spine Surgery and Research in the Region of Southern Denmark with symptomatic, MRI-verified lumbar spinal stenosis or disc herniations
* low risk (American Society of Anesthesiologists, ASA, score 1-2) adult patients scheduled for elective primary decompression or/and discectomy over one to two vertebral levels (without fusion or instrumentation), willing to give informed consent.

Exclusion Criteria:

Not able to understand verbal and/or written Danish ASA score more than 2 Malignant disease Pregnancy Breast feeding

Contraindications to TXA:

Active thromboembolic disease Coagulopathy History of venous or arterial thrombosis Hypersensitivity to the active substance Disseminated intravascular coagulation Severe renal impairment History of convulsions ASA - American Society of Anesthesiologists score, TXA - Tranexamic acid.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2016-08-16 (Actual); Study Completion 2016-08-16 (Actual)

PRIMARY OUTCOMES:
Operative time | Intraoperative (The time in minutes from incision to closure (last stitch) was measured)
  Defined as the time in minutes from incision to closure (last stitch)

SECONDARY OUTCOMES:
Perioperative bleeding and occurrence of dural tear, Deep venous thrombosis T. | Surgical drain volume was estimated visually at two and 18 hours post-operatively.
  Intra-operative blood loss was estimated by adding the weight (1g=1mL) of swabs and blood in the suction bottle and subtracting all fluids added to the surgical field. Surgical drain volume was estimated visually at two and 18 hours post-operatively. Total volume of peri-operative blood loss was calculated as the volume of intraoperative blood loss plus the post-operative volume measured from the drain output.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Andersen, MD, Study Chair — Sygehus Lillebaelt
Locations (1):
- Spine Center of Southern Denmark, Middelfart, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet, so no plan except publishing the result in a scientific paper.

REFERENCES:
- [Derived] Elmose S, Andersen MO, Andresen EB, Carreon LY. Double-blind, randomized controlled trial of tranexamic acid in minor lumbar spine surgery: no effect on operative time, intraoperative blood loss, or complications. J Neurosurg Spine. 2019 Apr 12;31(2):194-200. doi: 10.3171/2019.1.SPINE1814. Print 2019 Aug 1. PMID 30978683